CLINICAL TRIAL: NCT02908880
Title: Pivotal Clinical Study to EvaluAte the SaFety and Effectiveness of MANTA Vascular Closure Device
Brief Title: MANTA Percutaneous Vascular Closure Device - The SAFE MANTA Study
Acronym: SAFE_MANTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essential Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PSD-109
Record Dates: First submitted 2016-09-09; First posted 2016-09-21 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Femoral Arteriotomy Closure
Keywords: MANTA; Arterial Closure Device; Large Bore Closure Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MANTA vascular closure device (Experimental): Open label, single arm study using the MANTA device, developed by Essential Medical, Inc. MANTA is a vascular closure device (VCD) intended for use in catheterization laboratories following percutaneous cardiac or peripheral procedures that use the retrograde common femoral artery access route for large bore (10-18F) interventional devices.
  Interventions: Device: MANTA vascular closure device

INTERVENTIONS:
Device: MANTA vascular closure device — The appropriate size of MANTA closure device will be selected and used for the closure of femoral arterial access sites following the use of 10-14F devices or sheaths or the use of 15-18F devices or sheaths.
  Other Names: MANTA

SUMMARY:
Research study which tests the safety and effectiveness of a new vascular closure device to close the femoral access puncture that is created in patients who require this form of access in order to perform the planned procedure. The MANTA device is expected to seal the femoral access puncture in less than 1 minute. This may result in less blood loss and a shorter time to walking compared to alternative closure means. Use of the MANTA device in this study is experimental. All other parts of the procedure involve standard medical care.

DETAILED DESCRIPTION:
The MANTA device is a VCD intended for use in catheterization laboratories following percutaneous cardiac or peripheral procedures that use the retrograde common femoral artery access route for large bore (10-18F ID) interventional devices. The function of MANTA is to percutaneously close the puncture in the artery wall (arteriotomy) through which the catheters were inserted for the procedure.

The study is being conducted to demonstrate the safety and effectiveness of MANTA in achieving hemostasis in femoral arterial access sites in subjects undergoing percutaneous transcatheter interventional procedures using a large-bore procedure sheath.

ELIGIBILITY:
Inclusion Criteria:

1. Candidate for elective or planned (i.e., not emergent or urgent) percutaneous transcatheter interventional procedure via a 10-18F size retrograde common femoral artery approach (i.e., transcatheter aortic valve implantation [TAVI], endovascular aneurysm repair [EVAR], Impella® use)
2. Vessel size would allow for access for the MANTA device as determined by baseline CTA: minimum vessel diameter 5mm for the 14F MANTA and 6mm for the 18F MANTA
3. Eligible for sheath removal in the catheterization lab
4. Age ≥21 years
5. Understand and sign the study specific written informed consent form
6. Able and willing to fulfill the follow-up requirements
7. In the investigator's opinion, patient is suitable for the MANTA vascular closure device, conventional hemostasis techniques and participation in an investigational trial

Exclusion Criteria:

1. Known to be pregnant or lactating
2. Immunocompromised or with pre-existing autoimmune disease
3. Systemic infection or a local infection at or near the access site
4. Significant anemia (hemoglobin <10 g/DL, hematocrit <30%)
5. Morbidly obese or cachectic (BMI >40 kg/m2 or <20 kg/m2)
6. Known bleeding disorder including thrombocytopenia (platelet count <100,000 cells/UL), thrombasthenia, hemophilia, or von Willebrand disease
7. Allergy to bovine materials or any other device material, including collagen and/or collagen products, polyglycolic or polylactic acid, stainless steel or nickel
8. Femoral artery puncture in target groin within the prior 14 days
9. Previous iliofemoral intervention in region of access site, including but not limited to prior atherectomy, stenting, surgical or grafting procedures in the access area
10. Patients who have undergone use of an intra-aortic balloon pump through the arterial access site within 30 days prior to the baseline evaluation
11. Patients who are not mobile and are confined to a wheelchair or bed
12. NYHA class IV heart failure
13. Patients who have already participated in the IDE study
14. Currently participating in another clinical trial of an unapproved investigational device or drug that has not concluded the follow-up period
15. Patient cannot adhere to or complete the investigational protocol for any reason including but not limited to geographical residence, psychiatric condition or life threatening disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2016-12; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wood, MD, Principal Investigator — St. Paul's Hospital; Zvonimir Krajcer, MD, Principal Investigator — St. Luke's Episcopal
Locations (19):
- United States (18):
  - San Diego VA Medical Center, San Diego, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Evanston Hospital, Evanston, Illinois
  - St. Vincent Heart Center, Indianapolis, Indiana
  - Henry Ford, Detroit, Michigan
  - St. Luke Hospital (Mid America Heart), Kansas City, Missouri
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Lankenau Heart Group, Wynnewood, Pennsylvania
  - Avera Heart Hospital, Sioux Falls, South Dakota
  - Wellmont Holston Valley Hospital, Kingsport, Tennessee
  - Houston Methodist, Houston, Texas
  - St. Luke's Hospital - Texas Heart, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Swedish Medical Center, Seattle, Washington
  - CAMC Memorial Hospital, Charleston, West Virginia
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data obtained will be used, without mentioning Subject PHI, to assess the results of the research, and the data could be used in the future with regard to this study or other studies. The data can be passed on to the health authorities for the purposes of registering the medical device.

REFERENCES:
- [Derived] Krajcer Z, Wood DA, Strickman N, Bernardo N, Metzger C, Aziz M, Bacharach JM, Nanjundappa A, Campbell J, Lee JT, Dake MD, Lumsden A, Nardone S. Pivotal Clinical Study to Evaluate the Safety and Effectiveness of the MANTA Vascular Closure Device During Percutaneous EVAR and TEVAR Procedures. J Endovasc Ther. 2020 Jun;27(3):414-420. doi: 10.1177/1526602820912224. Epub 2020 Mar 20. PMID 32193971
- [Derived] Wood DA, Krajcer Z, Sathananthan J, Strickman N, Metzger C, Fearon W, Aziz M, Satler LF, Waksman R, Eng M, Kapadia S, Greenbaum A, Szerlip M, Heimansohn D, Sampson A, Coady P, Rodriguez R, Krishnaswamy A, Lee JT, Ben-Dor I, Moainie S, Kodali S, Chhatriwalla AK, Yadav P, O'Neill B, Kozak M, Bacharach JM, Feldman T, Guerrero M, Nanjundappa A, Bersin R, Zhang M, Potluri S, Barker C, Bernardo N, Lumsden A, Barleben A, Campbell J, Cohen DJ, Dake M, Brown D, Maor N, Nardone S, Lauck S, O'Neill WW, Webb JG; SAFE MANTA Study Investigators. Pivotal Clinical Study to Evaluate the Safety and Effectiveness of the MANTA Percutaneous Vascular Closure Device. Circ Cardiovasc Interv. 2019 Jul;12(7):e007258. doi: 10.1161/CIRCINTERVENTIONS.119.007258. Epub 2019 Jul 12. PMID 31296082

RESULTS

PARTICIPANT FLOW:
Groups:
- MANTA Vascular Closure Device: Open label, single arm study using the MANTA device, developed by Essential Medical, Inc.. MANTA is a vascular closure device (VCD) intended for use in catheterization laboratories following percutaneous cardiac or peripheral procedures that use the retrograde common femoral artery access route for large bore (10-18F) interventional devices.
  MANTA vascular closure device: The appropriate size of MANTA closure device will be selected and used to for the closure of femoral arterial access sites following the use of 10-14F devices or sheaths or the use of 15-18F devices or sheaths.
Period: Overall Study
Arm/Group | MANTA Vascular Closure Device
Started | 263 (Subjects within the Primary Analysis Cohort that received the MANTA Device)
Completed | 236 (Subjects within the Primary Analysis Cohort that completed all follow-up time points.)
Not Completed | 27
Not completed — Lost to Follow-up | 4
Not completed — Explantation of the device | 1
Not completed — Withdrawal by Subject | 17
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Arm/Group | MANTA Vascular Closure Device
Number analyzed (Participants) | 263
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.4 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 247
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 247
  More than one race | 0
  Unknown or Not Reported | 1
Ankle Brachial Index (ABI) [Mean (Standard Deviation); unit: ratio] | 1.1 (0.3)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (4.4)
Minimum Target Vessel Diameter [Mean (Standard Deviation); unit: mm] | 7.9 (1.4)
Creatinine [Mean (Standard Deviation); unit: umol/L] | 97.1 (27.7)
Hematocrit [Mean (Standard Deviation); unit: L/L] | 0.39 (0.04)
Hemoglobin [Mean (Standard Deviation); unit: mmol/L] | 8.1 (0.9)
Platelets [Mean (Standard Deviation); unit: 10^9/L] | 199.1 (63)

OUTCOME MEASURES:

1. Primary Outcome: Time to Hemostasis
Description: The elapsed time between withdrawal of MANTA sheath/device from artery and first observed and confirmed arterial hemostasis (no or minimal subcutaneous oozing and the absence of expanding or developing hematoma).
Time Frame: During access site closure, usually within an hour of starting the procedure.
Population: Primary Analysis Cohort
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | MANTA Vascular Closure Device
Number analyzed (Participants) | 263
seconds | 65.4 (157.8)

2. Primary Outcome: Number of Patients With Major Complications, Within 30 Days of Procedure
Description: IDE Protocol-Defined Major Complications analyzed on a per-patient basis
Time Frame: Up to 30 days after procedure
Population: Primary Analysis Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | MANTA Vascular Closure Device
Number analyzed (Participants) | 263
Participants | 14

3. Secondary Outcome: Technical Success
Description: Percutaneous vascular closure obtained with the MANTA device without the use of unplanned endovascular or surgical intervention
Time Frame: Within 6 hours after deployment of the MANTA device
Population: Primary Analysis Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | MANTA Vascular Closure Device
Number analyzed (Participants) | 263
Participants | 257

4. Secondary Outcome: Number of Patients With VARC-2 Major Vascular Complications, Adapted From the VARC-2 Criteria, Within 30 Days of Procedure
Description: Incidence of VARC-2 Major Vascular Complications, analyzed on a per-patient basis
Time Frame: Up to 30 days after procedure
Population: Primary Analysis Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | MANTA Vascular Closure Device
Number analyzed (Participants) | 263
Participants | 11

5. Secondary Outcome: Number of Patients With Minor Complications, Within 30 Days of Procedure
Description: Incidence of IDE Protocol-defined Minor Complications, analyzed on a per-patient analysis
Time Frame: Up to 30 days after procedure
Population: Primary Analysis Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | MANTA Vascular Closure Device
Number analyzed (Participants) | 263
Participants | 7

ADVERSE EVENTS:
Time Frame: Approximately 60 days after deployment of the MANTA device
Arm/Group | MANTA Vascular Closure Device
All-Cause Mortality (participants affected / at risk) | 5/263
Serious Adverse Events (participants affected / at risk) | 70/263
Other Adverse Events (participants affected / at risk) | 71/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MANTA Vascular Closure Device (N=263)
Anemia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Mild leukocytosis of non study leg (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 2
Complete Heart Block (Cardiac disorders) | 7
Pericardial effusion (Cardiac disorders) | 2
Heart Block (Cardiac disorders) | 4
Congestive Heart Failure Exacerbation (Cardiac disorders) | 5
Cardiogenic Shock (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 3
Left Bundle Branch Block (Cardiac disorders) | 2
Thrombus (Cardiac disorders) | 1
Sinus arrest (Cardiac disorders) | 1
AV Nodal Conduction Disorder (Cardiac disorders) | 1
Atrial Flutter (Cardiac disorders) | 1
Arrhythmia not otherwise noted (Cardiac disorders) | 1
Acute Cardiac Failure (Cardiac disorders) | 1
Severe Gastritis (Gastrointestinal disorders) | 1
Retroperitoneal bleed (Gastrointestinal disorders) | 2
Ischemic Bowel (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Fever (General disorders) | 2
Abnormal Gait (General disorders) | 1
Urinary Tract Infection (Infections and infestations) | 2
Septic Shock (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Systemic Infection (Infections and infestations) | 2
Access site bleeding-arterial (Injury, poisoning and procedural complications) | 1
Valve thrombosis or patient prothesis mismatch (Injury, poisoning and procedural complications) | 1
Pseudoaneurysm (Injury, poisoning and procedural complications) | 4
Access site Occlusion (Injury, poisoning and procedural complications) | 5
Multiple falls with prolonged immobilization (Injury, poisoning and procedural complications) | 1
Decrease in Ejection Fraction (Investigations) | 1
Local infection at location other than femoral access sites (Investigations) | 1
Acute gout on left knee (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
PPM pocket hematoma (Musculoskeletal and connective tissue disorders) | 1
Left arm and shoulder pain (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Recurrent lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vaso-vagal Event (Nervous system disorders) | 1
Acute Aphasia (Nervous system disorders) | 1
Stroke/cerebrovascular accident (Nervous system disorders) | 3
Intraparenchymal Hemorrhage in left frontal lobe (Nervous system disorders) | 1
Hemorrhage within horizontal sylvian fissure on left and intraventricular hemorrhage (Nervous system disorders) | 1
Acute Metabolic Encephalopathy (Nervous system disorders) | 1
Transient ischemic attack (Nervous system disorders) | 1
Decreased cardiac functional status (Product Issues) | 1
Acute urinary retention post TAVI (Renal and urinary disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 4
Acute Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1
Right lower lobe pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1
Femoral artery stenosis (Vascular disorders) | 2
Retrograde dissection originating at puncture site (Vascular disorders) | 1
Distal External Iliact Artery Stenosis >50% (Vascular disorders) | 1
Limb ischemia (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Hypovolemic shock (Vascular disorders) | 1
NSTEMI (Vascular disorders) | 1
Arterial embolism to limb (Vascular disorders) | 1
Type A Aortic dissection (Vascular disorders) | 2
Left Arm Hematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MANTA Vascular Closure Device (N=263)
Left Bundle Branch Block (Cardiac disorders) | 14
Access site bleeding-oozing (Injury, poisoning and procedural complications) | 39
Hematoma (Injury, poisoning and procedural complications) | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Typical language included: Research Institution and Principal Investigator agree that they shall not, without the Sponsor's prior written consent, independently Publish any results of or information about the activities conducted until the multi-center publication is released. If a multi-center manuscript is not submitted for publication within one (1) year after completion of the multi-center Study, Research Institution and Principal Investigator shall have the right to Publish results.

DOCUMENTS (2):
  • Study Protocol (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT02908880/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT02908880/SAP_001.pdf